CLINICAL TRIAL: NCT03947372
Title: Comparison of Outcomes After Laparoscopic Versus Open Appendectomy in Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Safia Zahir Ahmed, principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/451/SIMS
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Appendectomy; Pain, Postoperative; Length of Stay
Keywords: Open Appendectomy; Laparoscopic Appendectomy; post-operative pain; Hospital stay
MeSH Terms: conditions — Pain, Postoperative | interventions — Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA (open Appendectomy) (Active Comparator): Open Appendectomy
  Interventions: Procedure: Appendectomy
- LA (Laparoscopic Appendectomy) (Experimental): Laparoscopic Appendectomy
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — removal of acutely inflamed appendix

SUMMARY:
A comparison study was performed between laparoscopic appendectomy and open appendectomy in acute setting in tertiary hospital to access the outcome of postoperative pain and hospital stay. As the popularity of laparoscopic appendectomy has failed in major tertiary hospital due to huge amount of patient load in which open appendectomy was performed.This study was performed to prove that outcome of laparoscopic appendectomy are far better than open appendectomy and to increase the use of laparoscopic surgery in acute settings

DETAILED DESCRIPTION:
Introduction:

Open appendicectomy has been a safe and usually opted mode of operation for acute appendicitis for more than a century, but since last 10 years laparoscopic appendicectomy is gaining popularity, although still not as popular as laparoscopic cholecystectomy. Comparison of these two is studied in terms of pain outcome as patient perceives and length of hospital stay.

OBJECTIVES:

The objective of this study was to compare the outcome of open appendectomy and laparoscopic appendectomy in patients with acute appendicitis.

STUDY DESIGN: Randomized control trial

SETTING:

Surgical Unit I, Services Hospital, Lahore

DURATION OF STUDY:

Duration of my study was six months after the approval of synopsis i.e 21-02-2015 to 20-08-2015.

SAMPLE SIZE:

Was calculated using WHO method of calculating sample size.

SAMPLING TECHNIQUE:

Non probability consecutive sampling.

DATA COLLECTION PROCEDURE:

All patients fulfilled the inclusion criteria was admitted through the emergency after taking approval from hospital Ethical committee. A detailed history had been taken including demographic data (age, address). Patients was requested to sign an informed consent. They had been assured regarding confidentiality and expertise used for the procedure. All procedures was done by a single operating surgical team to control bias. All the data/variables was recorded on a specially designed Performa attached which are post-op pain at 12hrs and 24 hrs, post-Op stay and patient satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

* with acute appendicitis confirmed clinically by pain in right iliac fossa accompanied by right iliac fossa tenderness, elevated leukocyte count (>8*109/ml) without a palpable mass and on radiological investigation admitted through emergency department were included in the study.

Exclusion Criteria:

* • Perforated appendix (had been assesses on abdominal ultrasound or per-operatively.

  * Palpable mass in the right lower quadrant as assessed by clinical exam.
  * History of Co-morbidities e.g. known diabetic, known hypertensive, cirrhosis as shown by ultrasonography and coagulation disorder (to be determined by low platelet count; <140 *109, deranged PT and APTT).(PT=13sec, APTT= 33 sec)
  * Patients unfit for surgery (ASA Grade III/IV).
  * Patient who did not give informed consent.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2015-02-21 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Mean Post-operative pain | patient was assessed after 12 and 24 hours of surgery and change noted in 24 hour
  Visual Analogue Score at 12 and 24 hours after surgery . Score 0-10 where '0 shows no distress and '10' shows severe distress.
Hospital Stay | patient was assessed from 1 to 6 days after surgery
  Had been the total number of days spent in hospital during the same admission (from date of operation till date of discharge).Patient had been discharged as soon as bowel sounds are audible, passed flatus and resumed oral feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
share of Abstract and data to be shared on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: can be accessed on request